CLINICAL TRIAL: NCT04149717
Title: The Effect of Energy Drink Ingredients on Cardiovascular Function
Brief Title: The Effect of Energy Drink Ingredients on Cardiovascular Function in Men and Women 18-39 Years Old
Acronym: EEDICF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Duquesne University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: #2019/10/1
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2020-05

CONDITIONS: Cardiac Arrhythmia; Blood Pressure
Keywords: caffeine; taurine; carnitine; energy drink
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: repeated measures, crossover design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The three test solutions will be coded as "A", "B" and "C". Both the subject and the provider of the test solution to the subject will be blinded to the ingredients in the solution. The person who provides the test solution will be blind to the identity of the subject other than by subject number. The person who analyzes the data will be blinded to subject identity and which test solution was administered. The key for the test solutions and subject identity will be kept in a locked drawer in the office of the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Changes in BP, HR and EKG with Test Solution A and Exercise (Experimental): 1. Subject baseline HR, BP, EKG recorded.
  2. Subject will ingest sucrose (150g):
  3. 30 min later, subject will exercise on a treadmill
  4. Subjects will return each week to repeat the above procedures with a different test solution.
  Interventions: Dietary Supplement: Energy Drink Ingredients and Exercise
- Changes in BP, HR and EKG with Test Solution B and Exercise (Experimental): 1. Subject baseline HR, BP, ECG recorded.
  2. Subject will ingest sucrose (150g); caffeine (400 mg)
  3. 30 min later, subject will exercise on a treadmill
  4. Subjects will return each week to repeat the above procedures with a different test solution.
  Interventions: Dietary Supplement: Energy Drink Ingredients and Exercise
- Changes in BP, HR and EKG with Test Solution C and Exercise (Experimental): 1. Subject baseline HR, BP, ECG recorded.
  2. Subject will ingest sucrose (150g); caffeine (400 mg); taurine (4,000 mg); carnitine (400 mg)
  3. 30 min later, subject will exercise on a treadmill
  Interventions: Dietary Supplement: Energy Drink Ingredients and Exercise
- Changes in BP, HR and EKG with Test Solution C (Experimental): 1. Subject baseline HR, BP, ECG recorded.
  2. Subject will ingest sucrose (150g); caffeine (400 mg); taurine (4,000 mg); carnitine (400 mg)
  Interventions: Dietary Supplement: Energy Drink Ingredients and Exercise

INTERVENTIONS:
Dietary Supplement: Energy Drink Ingredients and Exercise — Subject will ingest 500 mL of one of three test solutions:
  A) sucrose (150g) B) sucrose (150g); caffeine (400 mg) C) sucrose (150g); caffeine (400 mg); taurine (4,000 mg); carnitine (400 mg) 3. 30 min later, subject will exercise on a treadmill using the Bruce Protocol maximum exercise test (https://www.aopa.org/go-fly/medical-resources/health-conditions/heart-and-circulatory-system/bru...). For one additional session, subjects will receive test solution C without exercise.
  4. Each stage will last 3 minutes. Stage 1 = 1.7 mph at 2% Grade Stage 2 = 2.5 mph at 4% Grade Stage 3 = 3.4 mph at 6% Grade Stage 4 = 4.2 mph at 8% Grade Stage 5 = 5.0 mph at 10% Grade Stage 6 = 5.5 mph at 12% Grade Stage 7 = 6.0 mph at 14% Grade Stage 8 = 6.5 mph at 15% Grade Stage 9 = 7.0 mph at 15% Grade. The test will end when subjects reach exhaustion.
  5. 1, 2, and 4 hrs following ingestion, HR, BP, and EKG will be recorded.

SUMMARY:
1. Statement of the research question:

   Does the caffeine in energy drinks interact with other ingredients to affect cardiovascular function in healthy male and female adults after exercise?
2. Purpose and significance of the study:

Energy drinks are beverages promoted to enhance alertness along with athletic and cognitive performance. The most common ingredients found in energy drinks include water, sugar, caffeine, taurine, and B-vitamins, with variable inclusion of other ingredients, such as carnitine, glucuronolactone, inositol, guarana, ginkgo biloba leaf extract, thistle extract, and ginseng root extract. Since the mid-1990s, the consumption of energy drinks has grown dramatically, with worldwide sales in 2017 exceeding $49 billion.

As the sale of energy drinks has grown, so has the number of adverse event case reports for patients who consumed energy drinks. Reported symptoms included cardiac arrhythmias such as ventricular fibrillation, atrial fibrillation, and cardiac arrest. A few small clinical studies have found that energy drinks can increase systolic and diastolic blood pressure and change electrical activity in the heart as measured by an electrocardiogram (ECG). The intent of the proposed study is to determine whether caffeine or the combination of caffeine with taurine and L-carnitine can alter cardiovascular function. Hypothesis: The effects of the ingredients of energy drinks on the heart are mediated in part by interactions between caffeine, taurine and carnitine. The amount of each ingredient in the study was based upon the amount commonly contained in two cans of energy drinks currently on the market.

DETAILED DESCRIPTION:
Title: The Effect of Energy Drink Ingredients on Cardiovascular Function

1. Statement of the research question

   Does the caffeine in energy drinks interact with other ingredients to affect cardiovascular function, including QTc interval of the EKG, heart rate and blood pressure in healthy male and female adults after exercise?
2. Purpose and significance of the study

Energy drinks are beverages promoted to enhance alertness along with athletic and cognitive performance. The most common ingredients found in energy drinks include water, sugar, caffeine, taurine, and B-vitamins, with variable inclusion of other ingredients, such as carnitine, glucuronolactone, inositol, guarana, ginkgo biloba leaf extract, thistle extract, and ginseng root extract. Since the mid-1990s, the consumption of energy drinks has grown dramatically, with worldwide sales in 2017 exceeding $49 billion.

As the sale of energy drinks has grown, so has the number of adverse event case reports for patients who consumed energy drinks. Reported symptoms include cardiac arrhythmias such as ventricular fibrillation, atrial fibrillation, and cardiac arrest. A few small clinical studies have reported that energy drinks can increase systolic and diastolic blood pressure and change electrical activity in the heart as measured by an electrocardiogram (EKG). The intent of the proposed study is to determine whether caffeine or the combination of caffeine with taurine and L-carnitine can alter heart rate, blood pressure and the QTc interval of the EKG. Caffeine stimulates cardiovascular function primarily through antagonism of adenosine receptors. Taurine is a modulator of intracellular calcium ion concentrations which can affect the strength cardiac contraction. Carnitine facilitates fatty acid transport into the mitochondria, thereby increasing the production of adenosine triphosphate, the energy source of cells. Hypothesis: the effects of the ingredients of energy drinks on the heart are mediated in part by interactions between caffeine, taurine and carnitine. The amount of each ingredient in the study was based upon the amount commonly contained in two cans of energy drinks currently on the market.

ELIGIBILITY:
Inclusion Criteria:

1. No preexisting medical conditions (including pregnancy)
2. Subjects must be capable of exercising on a treadmill (Vigorous activity: more than 7 kcal/min; https://www.cdc.gov/nccdphp/dnpa/physical/pdf/PA_Intensity_table_2_1.pdf)
3. BMI within normal range (18.5 - 24.9 kg/m2)
4. Average daily caffeine intake between 1 and 5 caffeinated beverages

Exclusion Criteria:

1. Age below 18 or greater than 39 years
2. Unable to provide legal consent to participate in the study
3. Preexisting medical conditions including but not limited to: pregnancy, cardiovascular disease, endocrine disorders, psychiatric or neurological disorders, musculo-skeletal disorders, immune disorders, respiratory disorders, dermatological disorders, infections, blindness, hearing disabilities
4. BMI less than 18.5 or greater than 24.9 kg/m25.
5. Current or future students of Drs. Johnson and/or Montepara
6. Incarceration in local, state or federal justice systems

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Change in QTc interval of EKG | 0, 1, 2, 4, hours post-dose
  Lengthening or shortening of the corrected QT interval (QTc) of the subject EKG at 1, 2, and 4 hours post treatment will be compared to pre-treatment measurements. The QTc will be calculated utilizing Bezett's formula.

SECONDARY OUTCOMES:
Change in Heart Rate | 0, 1, 2, 4, hours post-dose
  Increase or decrease in heart rate at 1, 2, and 4 hours post treatment compared to pre-treatment. Measurements of heart rate will be taken utilizing an automated sphygmomanometer
Change in Systolic and Diastolic Blood Pressure | 0, 1, 2, 4, hours post-dose
  Increase or decrease in systolic and diastolic blood pressure at 1, 2, and 4 hours post treatment compared to pre-treatment. Measurements of heart rate will be taken utilizing an automated sphygmomanometer.

CONTACTS AND LOCATIONS:
Overall Officials: David Delmonico, Ph.D., Study Chair — Institutional Review Board, Chair, Duquesne University
Locations (1):
- Duquesne University, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fletcher EA, Lacey CS, Aaron M, Kolasa M, Occiano A, Shah SA. Randomized Controlled Trial of High-Volume Energy Drink Versus Caffeine Consumption on ECG and Hemodynamic Parameters. J Am Heart Assoc. 2017 Apr 26;6(5):e004448. doi: 10.1161/JAHA.116.004448. PMID 28446495
- [Background] Kozik TM, Shah S, Bhattacharyya M, Franklin TT, Connolly TF, Chien W, Charos GS, Pelter MM. Cardiovascular responses to energy drinks in a healthy population: The C-energy study. Am J Emerg Med. 2016 Jul;34(7):1205-9. doi: 10.1016/j.ajem.2016.02.068. Epub 2016 Mar 2. PMID 27162113
- [Background] Goldfarb M, Tellier C, Thanassoulis G. Review of published cases of adverse cardiovascular events after ingestion of energy drinks. Am J Cardiol. 2014 Jan 1;113(1):168-72. doi: 10.1016/j.amjcard.2013.08.058. Epub 2013 Oct 4. PMID 24176062
- [Background] Shah SA, Szeto AH, Farewell R, Shek A, Fan D, Quach KN, Bhattacharyya M, Elmiari J, Chan W, O'Dell K, Nguyen N, McGaughey TJ, Nasir JM, Kaul S. Impact of High Volume Energy Drink Consumption on Electrocardiographic and Blood Pressure Parameters: A Randomized Trial. J Am Heart Assoc. 2019 Jun 4;8(11):e011318. doi: 10.1161/JAHA.118.011318. Epub 2019 May 29. PMID 31137991
- [Background] Longo N, Frigeni M, Pasquali M. Carnitine transport and fatty acid oxidation. Biochim Biophys Acta. 2016 Oct;1863(10):2422-35. doi: 10.1016/j.bbamcr.2016.01.023. Epub 2016 Jan 29. PMID 26828774
- [Background] Turnbull D, Rodricks JV, Mariano GF, Chowdhury F. Caffeine and cardiovascular health. Regul Toxicol Pharmacol. 2017 Oct;89:165-185. doi: 10.1016/j.yrtph.2017.07.025. Epub 2017 Jul 26. PMID 28756014
- [Background] Satoh H. Cardiac actions of taurine as a modulator of the ion channels. Adv Exp Med Biol. 1998;442:121-8. doi: 10.1007/978-1-4899-0117-0_16. PMID 9635023
- See also: Energy drink consumption frequency in the U.S. 2016, by age — https://www.statista.com/statistics/621710/energy-drink-consumption-frequency-in-the-us-by-age/
- See also: Energy Drink Sales — http://www.nutritionaloutlook.com/hero/614473
- See also: Bruce Protocol Stress Test — https://www.aopa.org/go-fly/medical-resources/health-conditions/heart-and-circulatory-system/bruce-protocol-stress-test